CLINICAL TRIAL: NCT05087498
Title: Effect of Autologous Cord Blood-mononuclear Cells Infusion on Immune Microenvironment in Infants Born Very Preterm in NICU: a Randomized Controlled Trial -The Premature Autologous Cord-blood Immunomodulatory Study (PAIRS)
Brief Title: Effect of Autologous Cord Blood-mononuclear Cells Infusion on Immune Microenvironment in Infants Born Very Preterm in NICU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yang jie, Professor, Guangdong Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Guangdong M CH
Record Dates: First submitted 2021-08-25; First posted 2021-10-21 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Immunomodulation Effect
Keywords: autologous cord blood mononuclear cells; monozygotic twins; very premature infants
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: eight pairs of VPMTs who were admitted to NICU to receive respiratory support right after birth. The infants were assigned (1:1) to receiving at least 2×107 ACB-MNCs/kg or normal saline, intravenously, within 24-h post-enrollment within each pair.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Once the enrollment was confirmed, the research physician contacted the research nurse. They were informed with the assignment and prepared the processed cord blood MNC or normal saline. After preparation, infusion bag was covered with shading bag and infused by light-blocking infusion tube, so that the nurses who conducted the infusion and all physicians who treated the baby were not aware of the treatment assignment. We used the code name of ACBMNC number 1 or number 2 to name the infusion fluid in the computerized physician order entry. The staff who collected and analyzed the patients' data and who followed up the patients were also blinded with the assignment. The research nurse and physician that knew the allocation of treatment did not make decisions in baby's clinical care. The parents or guardians were also not aware of the assignment. Therefore, this study was double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACBMNC infusion group (Experimental): Those assigned to the ACBMNC group will receive intravenous autologous cord blood mononuclear cells infusion within 24 h after process. Cell dose for all patients was 2-10×107 cells per kilogram.
  Interventions: Biological: autologous cord blood mononuclear cells
- control group (Placebo Comparator): Those in control group will receive an infusion of a placebo solution which is normal saline with the same volume per kg.
  Interventions: Biological: normal saline

INTERVENTIONS:
Biological: autologous cord blood mononuclear cells — preterm neonates less than 32 weeks are assigned to receive intravenous autologous cord blood mononuclear cells infusion (2-10×107cells/kg) within 24 hours after birth
  Arms: ACBMNC infusion group
Biological: normal saline — preterm neonates less than 32 weeks are assigned to receive normal saline within 24 hours after birth
  Arms: control group

SUMMARY:
Multi-omics (analysis of peripheral blood immune cells subset, peripheral blood MNCs transcriptome, soluble inflammatory cytokine profile in blood and airway secretion, lung and gut microbiota, and the interaction) analysis was used to profile immune alternation of infants with intravenous ACBMNC infusion in very preterm monozygotic twins

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, double-blinded trial involving eight pairs of VPMTs who were admitted to NICU to receive respiratory support right after birth. The infants were assigned (1:1) to receiving at least 2×107 ACB-MNCs/kg or normal saline, intravenously, within 24-h post-enrollment within each pair. Multi-omics (analysis of peripheral blood immune cells subset, peripheral blood MNCs transcriptome, soluble inflammatory cytokine profile in blood and airway secretion, lung and gut microbiota, and the interaction) analysis was used to profile immune alternation of infants with ACB-MNCs infusion, along with paired controls. Feasibility, safety and clinical outcomes improvement of the ACB-MNCs infusion in both short and long term were also assessed.

ELIGIBILITY:
Inclusion criteria

1. born at study hospitals;
2. monozygotic twins (confirmed by ultrasonographic diagnosis before birth and confirm again with obstetricians during and after delivery, as monochorionic diamniotic twins and monochorionic monoamniotic Twins twins were both monozygotic twins, therefore they will be both eligible);
3. gestational age (GA) <32 weeks (GA was calculated based on the date of the last menstrual period of the mother and an ultrasonographic screening performed during the first trimester of pregnancy);
4. enrolled within the first 24 postnatal hours;
5. free of severe perinatal asphyxia (defined as an Apgar score of 0-3 for more than 5 minutes, a cord blood gas pH <7.00, or both);
6. free of severe congenital anomalies or genetic syndromes;
7. free of maternal sepsis24,25;
8. Written informed consent is obtained from the parents or guardians of the infants;
9. Either of the twins has available umbilical cord blood (UCB) , and the cell number was no more than 10×107 cells per kilogram, but should not be less than 2×107 cells per kilogram.

Exclusion criteria

(1) they exhibit severe congenital abnormalities (detected via prenatal ultrasound); (2) expected to die within the first 24 hours; (3) diagnosed with severe twin-to-twin transfusion syndrome confirmed by prenatal ultrasonography24.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
immunomodulation effect | during 7 days after intervention
  analysis of peripheral blood immune cells subset, peripheral blood MNCs transcriptome, soluble inflammatory cytokine profile in blood and airway secretion, lung and gut microbiota, and the interaction
success rate of cord blood collection | during 6 months after intervention
  cord blood collection, cell available, infused cell number
complications | during 6 months after intervention
  frequency of complications such IVH, NEC, retinopathy of prematurity (ROP), respiratory distress syndrome (RDS), LOS, and persistent pulmonary hypertension of newborn (PPHN) and anemia.

OTHER OUTCOMES:
Duration of mechanical ventilation, oxygen therapy and hospitalization | 36 weeks of postmenstrual age or the discharge
  Duration of mechanical ventilation, oxygen therapy and hospitalization at 36 weeks of postmenstrual age or the discharge
the frequence of glucocorticoid, pulmonary surfactant, blood products and re-intubation | 36 weeks of postmenstrual age or the discharge
  the frequence of glucocorticoid, pulmonary surfactant, blood products and re-intubation at 36 weeks of postmenstrual age or the discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, Study Chair — Guangdong Women and Children Hospital
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
public
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: All time
Access Criteria: all

REFERENCES:
- [Derived] Zhuxiao R, Ruoyu H, Liling Y, Xuejun R, Chunhui Y, Wanfen R, Zhifeng C, Yiheng D, Qi Z, Wei W, Zhipeng L, Jingjun P, Qigai Y, Jie Y. Autologous cord blood mononuclear cell infusion for the prevention of bronchopulmonary dysplasia in very preterm monozygotic twins: A study protocol for a randomized, placebo-controlled, double-blinded multicenter trial. Front Pediatr. 2022 Dec 9;10:884366. doi: 10.3389/fped.2022.884366. eCollection 2022. PMID 36568414